CLINICAL TRIAL: NCT05660148
Title: Influence of Resentment and Forgivingness on Quality of Life in People Living With HIV
Acronym: FORGHIV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2022_843_0010
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Forgiveness; Hiv; Stress; Stigma; Health
Keywords: Forgiveness; forgivingness; Hiv; Stress; stigma; health
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Social Stigma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Life stress is strongly associated with poor mental and physical health and its effects explain significant morbidity and mortality. Forgiveness is one of the factors that can influence the effects of stress on health. By definition, forgiveness is the release of negative feelings, emotions, and behaviors - and possibly the release of positive feelings - toward an offender. Numerous studies have shown that forgiveness is associated with several mental and physical health benefits. The literature argues that high levels of propensity to forgive (trait) predispose that person to experience forgiveness (state) more often. In other words, a stronger forgiving disposition is believed to increase the experience of forgiveness, which, in turn, mitigates the negative effects of stress. Forgiveness is therefore a coping style that can play a beneficial role in the stress-health relationship. Patients living with HIV (PLHIV) are patients particularly exposed to stress, not only because of their chronic pathology but also because of the stigma attached to this disease. Very few studies have studied the impact of forgiveness (state or trait) on the physical health of PLHIV and even fewer the impact of an intervention promoting the disposition to forgive. The objective of this prospective observational monocentric study is to show in a very secular country that forgiveness has an effect on well-being as well as on other health parameters.

ELIGIBILITY:
Inclusion Criteria:

* Belonging to the PLHIV followed at the Amiens University Hospital, not likely to move within the year
* Possibility of follow-up in teleconsultation (usual support of the service)
* Benefiting from a social security scheme
* Consent to participate in the research

Exclusion Criteria:

* Erratic follow-up (non-compliance, predictable move) or moribund patient
* Illiterate or not speaking french

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients living with HIV (PLHIV) are patients particularly exposed to stress, not only because of their chronic pathology but also because of the stigma attached to this disease.Patients belonging to the PLHIV followed at the Amiens University Hospital, not likely to move within the year
Sampling Method: Non-Probability Sample
Enrollment: 206 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
establishment of correlation between the inclination to forgiveness and the quality of life | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No